CLINICAL TRIAL: NCT03622112
Title: A Phase 2b Randomised, Double Blind, Placebo-Controlled, Parallel Arm, Multi-Centre Study to Assess Efficacy and Safety of Multiple Dose Levels of AZD7594 DPI Given Once Daily for Twelve Weeks, Compared to Placebo, in Asthmatics Symptomatic on Low Dose ICS
Brief Title: A Study to Assess the Efficacy and Safety of Multiple Dose Levels of AZD7594 Administered Once Daily by Inhalation in Asthmatic Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D3741C00007
Record Dates: First submitted 2018-07-05; First posted 2018-08-09 (Actual); Results first posted 2020-11-27 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Asthma
Keywords: Inhaled non-steroidal glucocorticoid receptor modulator; Asthma; Inhaled corticosteroids.; Glucocorticoid receptor (GA) agonists.; Chronic obstructive pulmonary disease.; Short-acting B2 agonist.; Fluticasone furoate.
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: All double-blind medication kits will have similar appearance regardless of the IP (AZD7594 or placebo) contained in a DPI device and will be labelled using a unique medication identification number (Kit ID) that is linked to a treatment arm. IVRS/IWRS will assign the study medication to be dispensed to each subjects at Visit 3.
  Supplies of budesonide, FF and SABA (salbutamol/albuterol) will be open-label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- AZD7594 Dose 1 (Experimental): The randomized subjects will receive AZD7594 55 μg/50 μg (nominal/delivered dose), oral inhalation via dry powder inhaler (DPI) once daily.
  Interventions: Drug: AZD7594 DPI 55μg/50μg.
- AZD7594 Dose 2 (Experimental): The randomized subjects will receive AZD7594 99 µg/90 µg, oral inhalation via DPI once daily.
  Interventions: Drug: AZD7594 DPI 99 µg/90 µg
- AZD7594 Dose 3 (Experimental): The randomized subjects will receive treatment with AZD7594 198 µg/180 µg, oral inhalation via DPI once daily.
  Interventions: Drug: AZD7594 DPI 198 µg/180 µg
- AZD7594 Dose 4 (Experimental): The randomized subjects will receive treatment with AZD7594 396 µg/360 µg, oral inhalation via DPI once daily.
  Interventions: Drug: AZD7594 DPI 396 µg/360 µg once daily.
- AZD7594 Dose 5 (Experimental): The randomized subjects will receive treatment with AZD7594 792 µg/720 µg, oral inhalation via DPI once daily.
  Interventions: Drug: AZD7594 DPI 792 µg/720 µg
- Placebo (Placebo Comparator): The randomized subjects will receive AZD7594 matching placebo oral inhalation via DPI once daily.
  Interventions: Drug: Placebo for AZD7594 once daily.
- Fluticasone Furoate (Active Comparator): The randomized subjects will receive treatment with fluticasone furoate (FF) oral inhalation via DPI, 100 µg per nominal dose, once daily (open-label).
  Interventions: Drug: FF 100 µg once daily (open-label)

INTERVENTIONS:
Drug: AZD7594 DPI 55μg/50μg. — A non-steroidal and selective modulator of the GR.
  Arms: AZD7594 Dose 1
Drug: AZD7594 DPI 99 µg/90 µg — A non-steroidal and selective modulator of the GR.
  Arms: AZD7594 Dose 2
Drug: AZD7594 DPI 198 µg/180 µg — A non-steroidal and selective modulator of the GR.
  Arms: AZD7594 Dose 3
Drug: AZD7594 DPI 396 µg/360 µg once daily. — A non-steroidal and selective modulator of the GR.
  Arms: AZD7594 Dose 4
Drug: AZD7594 DPI 792 µg/720 µg — A non-steroidal and selective modulator of the GR.
  Arms: AZD7594 Dose 5
Drug: Placebo for AZD7594 once daily. — Placebo for AZD7594
  Arms: Placebo
Drug: FF 100 µg once daily (open-label) — Fluticasone furoate
  Arms: Fluticasone Furoate

SUMMARY:
This study will assess the efficacy and safety of multiple dose levels of AZD7594 administered once daily (QD) by inhalation in a 12-week treatment period on asthma subjects. The activity will be assessed by comparing AZD7594 to placebo. The comparison between active comparator (FF) and placebo will be used for bench marking. The efficacy is assessed by the evaluation of change in trough forced expiratory volume in 1 second (FEV1). The aim is to develop AZD7594 as a once daily inhaled non-steroidal selective GR modulator (SGRM), which may ultimately lead to better disease control of both chronic obstructive pulmonary disease (COPD) and asthma through improved efficacy and compliance. The overall rationale for developing a once daily AZD7594 in a dry powder inhaler (DPI) is to provide a safe and effective future treatment option for both asthma and COPD subjects.

DETAILED DESCRIPTION:
This is a randomised, placebo-controlled, double-blind multi center (8 countries: Europe, United States [US], South Africa, and Japan) study conducted on 714 subjects (102 subject per arm) with asthma symptomatic on low dose inhaled corticosteroids (ICS). The study consists of 3 periods:

* Run-in period (21-28 days; visits 1 to 3)
* Treatment period (12-week; Visits 4 to 7)
* Follow-up (1-week; visit 8).

The Run-in period consist of 3 visits: Screening visit (1), reversibility visit (2) and randomization visit (3). All subjects will sign an informed consent form (ICF) prior to participating in any study-specific procedures. Subjects found to be eligible at Visit 1 (Screening Visit) will discontinue all asthma medications and switch to low dose budesonide (200 μg twice a day [BID] in Europe and 180 μg BID in US) and rescue medication will be taken as needed. Subjects on long-acting beta agonist (LABA), fixed dose combination ICS/LABA treatment or a long-acting muscarinic antagonist (LAMA) will return for Visit 2 between 2 to 7 days after Visit 1 to have a sufficient wash-out time of their asthma medications. If reversibility criteria are met at Visit 2, subjects will proceed to Visit 3 (Randomization will occur within 21 to 28 days of Visit 1). At Visit 3, subjects who remain symptomatic while on low dose budesonide will be randomized in an overall ratio of 1:1:1:1:1:1:1 to one of 7 possible treatments and will receive inhalation powder via oral route:

* AZD7594 DPI 55μg [nominal strength]/50 μg [delivered dose] (QD)
* AZD7594 DPI 99 μg/90 μg QD
* AZD7594 DPI 198 μg/180 μg QD
* AZD7594 DPI 396 μg/360 μg QD
* AZD7594 DPI 792 μg/720 μg QD
* Placebo for AZD7594 QD
* FF 100 μg QD (open-label) The follow-up will be done by telephone contact within 7 to 10 days after Visit 7 or last investigational product (IP) intake.

The total duration of the study will be between 113 to 135 days for each individual subject and is planned to run approximately 12 months (it should not exceed 18 months).

ELIGIBILITY:
Inclusion criteria

1. Provision of informed consent prior to any study-specific procedures 2. Men and women 18 to 85 years of age, inclusive, with body mass index (BMI)≤35 3. Subjects need to be non-smokers or ex-smokers (have quit e cigarettes or other inhaled tobacco products ≥6 months before Visit 1) with a total smoking history of less than 10 pack-years (not applicable for e cigarettes) 4. Documented clinical diagnosis of asthma for ≥6 months before Visit 1 5. Subjects on stable medium to high dose ICS (equivalent of budesonide >400 μg/day) or low to medium dose ICS/LABA for at least 4 weeks prior to screening (Visit 1) (Appendix A, GINA, 2018) 6. Subjects must demonstrate reversibility to inhaled bronchodilators at Visit 2 (a ≥12% and ≥200 mL improvement in FEV1 after administration of a 4 puffs of salbutamol/albuterol) 7. Pre-bronchodilator FEV1 at Visit 3 between 40% and 90% predicted at either -45 or -15 minutes pre-dose 8. At Visit 3, subjects need to be symptomatic on low dose ICS as evidenced by combined daily asthma mean symptom score of >1 over the previous 7 days or SABA use on ≥3 of the last 7 days during the Run-in Period 9. Demonstrate the ability to use the study inhalation device properly 10. Subject able to perform acceptable pulmonary function testing for FEV1 according to American Thoracic Society/European Respiratory Society (ATS/ERS) acceptability criteria 11. Subject is willing and able to follow study procedures and restrictions. Women of child bearing potential (WOCBP) should be stable on their chosen method of highly effective birth control for a minimum of 3 months prior to Visit 1, and willing to use that for the entire duration of the study (from the time they sign the informed consent), and for 1 month after the last dose of IP 12. For optional inclusion in the Gx component of the study, subjects must provide separate informed consent for the genomic sampling and analysis Exclusion criteria

1. Known or suspected hypersensitivity to any of the IPs, including budesonide, or excipients, including lactose
2. Systemic steroid use within the 6 weeks before Visit 1
3. Concomitant chronic respiratory disease (including current sleep apnea)
4. History or clinical suspicion of any clinically relevant or active disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study, or any other safety concerns in the opinion of the Investigator
5. Use of prohibited medications that cannot be stopped during the entire period of the study (starting Visit 1).
6. Subjects with <80% eDiary compliance during Run in Period at Visit 3
7. ACQ-5 of ≥3 at Visit 1, Visit 2, or Visit 3
8. Daily rescue use of SABA ≥12 puffs for ≥3 consecutive days at any time during Run-in Period, before randomisation
9. Any clinically important abnormalities in rhythm, conduction or morphology of the digital ECG at rest and any abnormalities in the digital ECG (at Visit 1 or Visit 3) that, as considered by the Investigator, may interfere with the interpretation of QT interval corrected (QTc) interval changes
10. Prolonged QT interval corrected using Fridericia's formula (QTcF) ≥450 msec based on ECG at Visit 1 or Visit 3; or family history of long QT syndrome
11. PR (PQ) interval prolongation (>240 msec), intermittent second or third degree atrial-ventricular (AV) block or AV dissociation at Visit 1 or Visit 3
12. Subjects with implantable cardiac defibrillator and subjects with sustained symptomatic ventricular and/or atrial tachyarrhythmia
13. Subjects with unstable angina pectoris or stable angina pectoris classified higher than Canadian Cardiovascular Society Class II, or a myocardial infarction or stroke within 6 months before Visit 1
14. History of hospitalisation within 12 months before Visit 1 caused by heart failure or a diagnosis of heart failure higher than New York Heart Association Class II
15. Subjects who are positive for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody or human immunodeficiency virus (HIV) at Visit 1
16. Donation of blood (≥ 450 mL) within 3 months or donation of plasma within 14 days before Visit 1
17. Suspected poor capability to follow instructions of the study, as judged by the Investigator
18. Previous participation or prior screen failure in the current study, or participation in any other research study within 1 month prior to Visit 1
19. Subject under treatment with biologicals such as monoclonal antibodies or chimeric biomolecules including omalizumab, mepolizumab, and reslizumab within 6 months or 5 half-lives before Visit 1, whichever is longer
20. Subject treated with any investigational drug within 30 days (or 5 half-lives, whichever is longer) prior to Visit 1
21. Positive drug screening result that cannot be justified by subject's medical history and its relevant treatment (over-the-counter product or a valid prescription), or history of or current alcohol or drug abuse (including marijuana and marijuana-containing valid prescriptions), as judged by the Investigator
22. Planned in-patient surgery, major dental procedure or hospitalisation during the study
23. Pregnant woman or lactating woman
24. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff, contract research organisation staff and/or staff at the study centre)
25. Suspicion of Gilbert's syndrome
26. Vulnerable persons (eg, persons kept in detention)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 808 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kai Michael Beeh, Dr med, Principal Investigator — Insaf - Institut für Atemwegsforschung GmbH, D65187, Germany.
Locations (83):
- United States (21):
  - Research Site, Sheffield, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Fullerton, California
  - Research Site, Gold River, California
  - Research Site, New Haven, Connecticut
  - Research Site, Celebration, Florida
  - Research Site, Miami, Florida
  - Research Site, Port Orange, Florida
  - Research Site, Winter Park, Florida
  - Research Site, North Dartmouth, Massachusetts
  - Research Site, Farmington Hills, Michigan
  - Research Site, Charlotte, North Carolina
  - Research Site, Gastonia, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Dublin, Ohio
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Spartanburg, South Carolina
  - Research Site, Boerne, Texas
  - Research Site, San Antonio, Texas
- Bulgaria (7):
  - Research Site, Gabrovo
  - Research Site, Kozloduy
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Stara Zagora
  - Research Site, Vidin
- Germany (8):
  - Research Site, Berlin
  - Research Site, Dortmund
  - Research Site, Großhansdorf
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Lübeck
  - Research Site, Marburg
  - Research Site, Wiesbaden
- Hungary (10):
  - Research Site, Balassagyarmat
  - Research Site, Budapest
  - Research Site, Gödöllő
  - Research Site, Komló
  - Research Site, Miskolc
  - Research Site, Nyíregyháza
  - Research Site, Pécs
  - Research Site, Százhalombatta
  - Research Site, Szigetszentmiklós
  - Research Site, Szombathely
- Japan (12):
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Himeji
  - Research Site, Kagoshima
  - Research Site, Kishiwada-shi
  - Research Site, Naka-gun
  - Research Site, Osaka
  - Research Site, Sakaide-shi
  - Research Site, Shinjuku-ku
  - Research Site, Tokyo
  - Research Site, Yanagawa-shi
  - Research Site, Yokohama
- Poland (11):
  - Research Site, Bialystok
  - Research Site, Częstochowa
  - Research Site, Kielce
  - Research Site, Krakow
  - Research Site, Ksawerów
  - Research Site, Ostrowiec Świętokrzyski
  - Research Site, Proszowice
  - Research Site, Skarżysko-Kamienna
  - Research Site, Skierniewice
  - Research Site, Sopot
  - Research Site, Tarnów
- South Africa (4):
  - Research Site, Bellville
  - Research Site, Johannesburg
  - Research Site, Mowbray
  - Research Site, Port Elizabeth
- Ukraine (10):
  - Research Site, Cherkasy
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv Region
  - Research Site, Kyiv
  - Research Site, Lutsk
  - Research Site, Odesa
  - Research Site, Poltava
  - Research Site, Sumy
  - Research Site, Vinnytsia
  - Research Site, Zaporizhzhia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The CSP redacted. — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3741C00007&attachmentIdentifier=5b282157-6140-4ffe-a6f6-097cdf06eb7d&fileName=238537_English_Protocol_v2.0_Final_21-Sep-2020_Redacted.pdf&versionIdentifier=
- See also: The SAP redacted. — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3741C00007&attachmentIdentifier=c7bd3eb3-a5e0-4042-99df-402945d8f72d&fileName=238537_SAP_20191108_v3.0_Final_21-Sep-2020_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 92 sites in 8 countries; Bulgaria, Germany, Hungary, Poland, and Ukraine, United States (US), South Africa, and Japan. In this study, 806 patients (including 82 Japanese patients) were randomised. For sites in the US, no patients were randomised to the AZD7594 792 μg/720 μg once daily (QD) treatment arm.
Pre-assignment Details: Subjects attended a Screening Visit within 28 days before receiving their first dose. All subjects underwent inclusion exclusion criteria assessment and all eligible subjects signed the informed consent before undergoing any study related procedures. One patient in the AZD7594 50 μg treatment arm did not receive any treatment and was randomised in error (protocol deviation).
Groups:
- AZD7594 50 μg: Oral inhalation of AZD5794 55 microgram/ 50 microgram (nominal dose/delivered dose) once daily.
- AZD7594 90 μg: Oral inhalation of AZD5794 99 microgram/ 90 microgram (nominal dose/delivered dose) once daily.
- AZD7594 180 μg: Oral inhalation of AZD5794 198 microgram/ 180 microgram (nominal dose/delivered dose) once daily.
- AZD7594 360 μg: Oral inhalation of AZD5794 396 microgram/ 360 microgram (nominal dose/delivered dose) once daily.
- AZD7594 720 μg: Oral inhalation of AZD5794 792 microgram/ 720 microgram (nominal dose/delivered dose) once daily.
- Placebo to AZD7594: Oral inhalation of placebo to AZD7594 once daily.
- Fluticasone Furoate: Oral inhalation of fluticasone furoate 100 microgram once daily.
Period: Overall Study
Arm/Group | AZD7594 50 μg | AZD7594 90 μg | AZD7594 180 μg | AZD7594 360 μg | AZD7594 720 μg | Placebo to AZD7594 | Fluticasone Furoate
Started (One patient in the AZD7594 50 μg treatment arm did not receive any treatment and was randomised in error (protocol deviation).) | 110 | 112 | 111 | 113 | 134 | 113 | 112
Completed | 85 | 92 | 95 | 91 | 124 | 71 | 103
Not Completed | 25 | 20 | 16 | 22 | 10 | 42 | 9
Not completed — Withdrawal by Subject | 6 | 2 | 4 | 2 | 1 | 2 | 2
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Study-specific withdrawal criteria | 10 | 8 | 7 | 6 | 4 | 18 | 4
Not completed — Protocol Violation | 2 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 6 | 8 | 4 | 11 | 4 | 20 | 2
Not completed — Reason not specified | 0 | 1 | 0 | 1 | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD7594 50 μg | AZD7594 90 μg | AZD7594 180 μg | AZD7594 360 μg | AZD7594 720 μg | Placebo to AZD7594 | Fluticasone Furoate | Total
Number analyzed (Participants) | 110 | 112 | 111 | 113 | 134 | 113 | 112 | 805
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 90 | 92 | 79 | 92 | 107 | 87 | 82 | 629
  >=65 years | 20 | 20 | 32 | 21 | 27 | 26 | 30 | 176
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.2 (12.8) | 53.2 (13.3) | 54.6 (14.5) | 52.8 (13.2) | 52.2 (13.0) | 53.4 (13.7) | 53.7 (13.4) | 53.1 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 66 | 72 | 64 | 79 | 68 | 59 | 467
  Male | 51 | 46 | 39 | 49 | 55 | 45 | 53 | 338
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 9 | 11 | 10 | 13 | 16 | 13 | 12 | 84
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 5 | 5 | 2 | 1 | 5 | 7 | 30
  White | 95 | 93 | 94 | 97 | 115 | 92 | 93 | 679
  More than one race | 1 | 2 | 2 | 1 | 2 | 3 | 0 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough FEV1 at Week 12
Description: Trough value was defined as the mean of the 2 measurements 30 minutes apart (23 hours after last dose) pre-dose for every visit throughout the Treatment Period (Visit 4/Week 2 to Visit 7/Week 12). Baseline was defined as the mean of the 2 measured values before first IP administration (30 minutes apart, at -45 minutes and -15 minutes, before IP administration) on Day 1 (Visit 3). Analyses were based on a Mixed-effects model for repeated measures (MMRM) with treatment, visit, treatment by visit interaction and region as fixed effects, and baseline value and baseline by visit interaction as covariates. To investigate the clinical efficacy of AZD7594 at different dose levels in asthmatics symptomatic on low dose Inhaled corticosteroid (ICS).
Time Frame: At week 12
Population: Full Analysis Set: All participants randomised and receiving at least 1 dose of randomised study drug.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | AZD7594 50 μg | AZD7594 90 μg | AZD7594 180 μg | AZD7594 360 μg | AZD7594 720 μg | Placebo to AZD7594 | Fluticasone Furoate
Number analyzed (Participants) | 110 | 112 | 111 | 113 | 134 | 113 | 112
Liters | -0.013 [-0.077 to 0.050] | -0.031 [-0.094 to 0.031] | 0.062 [-0.001 to 0.124] | 0.099 [0.036 to 0.161] | 0.104 [0.046 to 0.162] | 0.022 [-0.046 to 0.091] | 0.133 [0.073 to 0.193]
Statistical Analysis 1: Comparison: AZD7594 50 μg vs Placebo to AZD7594; Test type: Superiority; p = 0.437, Mixed Models Analysis; Mean Difference (Final Values) = -0.036, 95% CI 2-sided [-0.126 to 0.054]
Statistical Analysis 2: Comparison: AZD7594 90 μg vs Placebo to AZD7594; Test type: Superiority; p = 0.236, Mixed Models Analysis; Mean Difference (Final Values) = -0.054, 95% CI 2-sided [-0.143 to 0.035]
Statistical Analysis 3: Comparison: AZD7594 180 μg vs Placebo to AZD7594; Test type: Superiority; p = 0.389, Mixed Models Analysis; Mean Difference (Final Values) = 0.039, 95% CI 2-sided [-0.050 to 0.128]
Statistical Analysis 4: Comparison: AZD7594 360 μg vs Placebo to AZD7594; Test type: Superiority; p = 0.094, Mixed Models Analysis; Mean Difference (Final Values) = 0.076, 95% CI 2-sided [-0.013 to 0.165]
Statistical Analysis 5: Comparison: AZD7594 720 μg vs Placebo to AZD7594; Test type: Superiority; p = 0.060, Mixed Models Analysis; Mean Difference (Final Values) = 0.082, 95% CI 2-sided [-0.003 to 0.167]
Statistical Analysis 6: Comparison: Placebo to AZD7594 vs Fluticasone Furoate; Test type: Superiority; p = 0.014, Mixed Models Analysis; Mean Difference (Final Values) = 0.111, 95% CI 2-sided [0.023 to 0.199]

2. Secondary Outcome: Change From Baseline in Trough FEV1 at Weeks 2, 4, 8 and Average Over the Treatment Period
Description: Trough value was defined as the mean of the 2 measurements 30 minutes apart (23 hours after last dose) pre-dose for every visit throughout the Treatment Period (Visit 4/Week 2 to Visit 7/Week 12). Baseline was defined as the mean of the 2 measured values before first IP administration (30 minutes apart, at -45 minutes and -15 minutes, before IP administration) on Day 1 (Visit 3). Analysis of covariance (ANCOVA) with treatment and region (ie, US, Japan, and RoW) as fixed effects, and baseline as covariate was used for the analysis of average over the Treatment Period. To investigate the clinical efficacy of AZD7594 at different dose levels in asthmatics symptomatic on low dose ICS.
Time Frame: At week 2, 4 and 8
Population: Full analysis set: All participants randomised and receiving at least 1 dose of randomised study drug.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | AZD7594 50 μg | AZD7594 90 μg | AZD7594 180 μg | AZD7594 360 μg | AZD7594 720 μg | Placebo to AZD7594 | Fluticasone Furoate
Number analyzed (Participants) | 110 | 112 | 111 | 113 | 134 | 113 | 112
Liters
  Week 2: number analyzed (Participants) | 108 | 107 | 108 | 104 | 132 | 95 | 109
  Week 2 | 0.018 [-0.038 to 0.073] | 0.011 [-0.044 to 0.066] | 0.067 [0.011 to 0.122] | 0.091 [0.036 to 0.147] | 0.093 [0.041 to 0.146] | -0.011 [-0.070 to 0.048] | 0.107 [0.052 to 0.161]
  Week 4: number analyzed (Participants) | 98 | 103 | 103 | 104 | 127 | 84 | 110
  Week 4 | -0.002 [-0.063 to 0.059] | 0.039 [-0.021 to 0.099] | 0.078 [0.018 to 0.138] | 0.086 [0.027 to 0.146] | 0.094 [0.037 to 0.151] | -0.020 [-0.085 to 0.045] | 0.145 [0.086 to 0.204]
  Week 8: number analyzed (Participants) | 90 | 96 | 100 | 96 | 125 | 76 | 105
  Week 8 | 0.019 [-0.044 to 0.082] | 0.007 [-0.055 to 0.069] | 0.071 [0.010 to 0.133] | 0.102 [0.040 to 0.163] | 0.141 [0.083 to 0.199] | 0.002 [-0.066 to 0.069] | 0.124 [0.064 to 0.184]
  Treatment Period Avg: number analyzed (Participants) | 108 | 109 | 108 | 109 | 132 | 95 | 110
  Treatment Period Avg | 0.005 [-0.049 to 0.059] | 0.006 [-0.047 to 0.059] | 0.069 [0.016 to 0.123] | 0.094 [0.041 to 0.148] | 0.108 [0.057 to 0.159] | -0.002 [-0.059 to 0.056] | 0.127 [0.075 to 0.180]
Statistical Analysis 1: Comparison: AZD7594 50 μg vs Placebo to AZD7594; Week 2; Test type: Superiority; p = 0.463, Mixed Models Analysis; Mean Difference (Final Values) = 0.029, 95% CI 2-sided [-0.048 to 0.105]
Statistical Analysis 2: Comparison: AZD7594 90 μg vs Placebo to AZD7594; Week 2; Test type: Superiority; p = 0.576, Mixed Models Analysis; Mean Difference (Final Values) = 0.022, 95% CI 2-sided [-0.055 to 0.098]
Statistical Analysis 3: Comparison: AZD7594 180 μg vs Placebo to AZD7594; Week 2; Test type: Superiority; p = 0.047, Mixed Models Analysis; Mean Difference (Final Values) = 0.078, 95% CI 2-sided [0.001 to 0.154]
Statistical Analysis 4: Comparison: AZD7594 360 μg vs Placebo to AZD7594; Week 2; Test type: Superiority; p = 0.009, Mixed Models Analysis; Mean Difference (Final Values) = 0.102, 95% CI 2-sided [0.025 to 0.179]
Statistical Analysis 5: Comparison: AZD7594 720 μg vs Placebo to AZD7594; Week 2; Test type: Superiority; p = 0.006, Mixed Models Analysis; Mean Difference (Final Values) = 0.104, 95% CI 2-sided [0.031 to 0.178]
Statistical Analysis 6: Comparison: Placebo to AZD7594 vs Fluticasone Furoate; Week 2; Test type: Superiority; p = 0.003, Mixed Models Analysis; Mean Difference (Final Values) = 0.118, 95% CI 2-sided [0.041 to 0.194]
Statistical Analysis 7: Comparison: AZD7594 50 μg vs Placebo to AZD7594; Week 4; Test type: Superiority; p = 0.685, Mixed Models Analysis; Mean Difference (Final Values) = 0.018, 95% CI 2-sided [-0.068 to 0.103]
Statistical Analysis 8: Comparison: AZD7594 90 μg vs Placebo to AZD7594; Week 4; Test type: Superiority; p = 0.176, Mixed Models Analysis; Mean Difference (Final Values) = 0.059, 95% CI 2-sided [-0.026 to 0.144]
Statistical Analysis 9: Comparison: AZD7594 180 μg vs Placebo to AZD7594; Week 4; Test type: Superiority; p = 0.024, Mixed Models Analysis; Mean Difference (Final Values) = 0.098, 95% CI 2-sided [0.013 to 0.183]
Statistical Analysis 10: Comparison: AZD7594 360 μg vs Placebo to AZD7594; Week 4; Test type: Superiority; p = 0.014, Mixed Models Analysis; Mean Difference (Final Values) = 0.106, 95% CI 2-sided [0.021 to 0.191]
Statistical Analysis 11: Comparison: AZD7594 720 μg vs Placebo to AZD7594; Week 4; Test type: Superiority; p = 0.006, Mixed Models Analysis; Mean Difference (Final Values) = 0.114, 95% CI 2-sided [0.032 to 0.196]
Statistical Analysis 12: Comparison: Placebo to AZD7594 vs Fluticasone Furoate; Week 4; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.165, 95% CI 2-sided [0.081 to 0.249]
Statistical Analysis 13: Comparison: AZD7594 50 μg vs Placebo to AZD7594; Week 8; Test type: Superiority; p = 0.707, Mixed Models Analysis; Mean Difference (Final Values) = 0.017, 95% CI 2-sided [-0.072 to 0.106]
Statistical Analysis 14: Comparison: AZD7594 90 μg vs Placebo to AZD7594; Week 8; Test type: Superiority; p = 0.904, Mixed Models Analysis; Mean Difference (Final Values) = 0.005, 95% CI 2-sided [-0.083 to 0.094]
Statistical Analysis 15: Comparison: AZD7594 180 μg vs Placebo to AZD7594; Week 8; Test type: Superiority; p = 0.121, Mixed Models Analysis; Mean Difference (Final Values) = 0.070, 95% CI 2-sided [-0.018 to 0.157]
Statistical Analysis 16: Comparison: AZD7594 360 μg vs Placebo to AZD7594; Week 8; Test type: Superiority; p = 0.026, Mixed Models Analysis; Mean Difference (Final Values) = 0.100, 95% CI 2-sided [0.012 to 0.188]
Statistical Analysis 17: Comparison: AZD7594 720 μg vs Placebo to AZD7594; Week 8; Test type: Superiority; p = 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.139, 95% CI 2-sided [0.055 to 0.224]
Statistical Analysis 18: Comparison: Placebo to AZD7594 vs Fluticasone Furoate; Week 8; Test type: Superiority; p = 0.006, Mixed Models Analysis; Mean Difference (Final Values) = 0.122, 95% CI 2-sided [0.035 to 0.209]
Statistical Analysis 19: Comparison: AZD7594 50 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.856, Mixed Models Analysis; Mean Difference (Final Values) = 0.007, 95% CI 2-sided [-0.068 to 0.081]
Statistical Analysis 20: Comparison: AZD7594 90 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.832, Mixed Models Analysis; Mean Difference (Final Values) = 0.008, 95% CI 2-sided [-0.066 to 0.082]
Statistical Analysis 21: Comparison: AZD7594 180 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.060, Mixed Models Analysis; Mean Difference (Final Values) = 0.071, 95% CI 2-sided [-0.003 to 0.145]
Statistical Analysis 22: Comparison: AZD7594 360 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.011, Mixed Models Analysis; Mean Difference (Final Values) = 0.096, 95% CI 2-sided [0.022 to 0.170]
Statistical Analysis 23: Comparison: AZD7594 720 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.003, Mixed Models Analysis; Mean Difference (Final Values) = 0.110, 95% CI 2-sided [0.039 to 0.181]
Statistical Analysis 24: Comparison: Placebo to AZD7594 vs Fluticasone Furoate; Treatment period average; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.129, 95% CI 2-sided [0.055 to 0.202]

3. Secondary Outcome: Change From Baseline in Fractional Exhaled Nitic Oxide (FENO) at Weeks 2, 4, 8, 12 and Average Over the Treatment Period
Description: Baseline was defined as the last value obtained prior to the first dose of investigational product. Analyses were based on a MMRM with change from baseline on the log-scale as the response, treatment, visit, treatment by visit interaction and region as fixed effects, and log-transformed baseline value and baseline by visit interaction as covariates.
Time Frame: At week 2, 4, 8, and 12
Population: Full Analysis Set: All participants randomised and receiving at least 1 dose of randomised study drug.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ppb
Arm/Group | AZD7594 50 μg | AZD7594 90 μg | AZD7594 180 μg | AZD7594 360 μg | AZD7594 720 μg | Placebo to AZD7594 | Fluticasone Furoate
Number analyzed (Participants) | 110 | 112 | 111 | 113 | 134 | 113 | 112
ppb
  Week 2: number analyzed (Participants) | 107 | 105 | 107 | 102 | 127 | 95 | 104
  Week 2 | 1.307 [1.190 to 1.436] | 1.223 [1.113 to 1.343] | 1.175 [1.070 to 1.290] | 1.152 [1.048 to 1.267] | 0.959 [0.876 to 1.049] | 1.396 [1.263 to 1.542] | 0.880 [0.801 to 0.967]
  Week 4: number analyzed (Participants) | 95 | 100 | 103 | 102 | 126 | 84 | 105
  Week 4 | 1.229 [1.109 to 1.363] | 1.203 [1.087 to 1.332] | 1.220 [1.103 to 1.349] | 1.118 [1.011 to 1.237] | 0.980 [0.891 to 1.078] | 1.321 [1.184 to 1.475] | 0.928 [0.840 to 1.025]
  Week 8: number analyzed (Participants) | 87 | 90 | 97 | 93 | 122 | 76 | 101
  Week 8 | 1.294 [1.157 to 1.447] | 1.316 [1.179 to 1.470] | 1.250 [1.122 to 1.392] | 1.206 [1.082 to 1.345] | 1.021 [0.923 to 1.129] | 1.411 [1.252 to 1.591] | 0.906 [0.815 to 1.007]
  Week 12: number analyzed (Participants) | 79 | 89 | 89 | 88 | 121 | 70 | 100
  Week 12 | 1.367 [1.219 to 1.532] | 1.405 [1.258 to 1.569] | 1.281 [1.148 to 1.431] | 1.198 [1.072 to 1.337] | 0.958 [0.866 to 1.060] | 1.474 [1.305 to 1.664] | 0.918 [0.826 to 1.022]
  Treatment Period Avg: number analyzed (Participants) | 109 | 107 | 108 | 109 | 132 | 95 | 110
  Treatment Period Avg | 1.298 [1.188 to 1.419] | 1.284 [1.176 to 1.402] | 1.231 [1.128 to 1.343] | 1.168 [1.070 to 1.275] | 0.979 [0.901 to 1.064] | 1.399 [1.273 to 1.538] | 0.908 [0.833 to 0.989]
Statistical Analysis 1: Comparison: AZD7594 50 μg vs Placebo to AZD7594; Week 2; Test type: Superiority; p = 0.322, Mixed Models Analysis; Mean Difference (Final Values) = 0.936, 95% CI 2-sided [0.822 to 1.067]
Statistical Analysis 2: Comparison: AZD7594 90 μg vs Placebo to AZD7594; Week 2; Test type: Superiority; p = 0.047, Mixed Models Analysis; Mean Difference (Final Values) = 0.876, 95% CI 2-sided [0.768 to 0.999]
Statistical Analysis 3: Comparison: AZD7594 180 μg vs Placebo to AZD7594; Week 2; Test type: Superiority; p = 0.010, Mixed Models Analysis; Mean Difference (Final Values) = 0.842, 95% CI 2-sided [0.739 to 0.959]
Statistical Analysis 4: Comparison: AZD7594 360 μg vs Placebo to AZD7594; Week 2; Test type: Superiority; p = 0.004, Mixed Models Analysis; Mean Difference (Final Values) = 0.825, 95% CI 2-sided [0.724 to 0.941]
Statistical Analysis 5: Comparison: AZD7594 720 μg vs Placebo to AZD7594; Week 2; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.687, 95% CI 2-sided [0.606 to 0.779]
Statistical Analysis 6: Comparison: Placebo to AZD7594 vs Fluticasone Furoate; Week 2; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.630, 95% CI 2-sided [0.553 to 0.719]
Statistical Analysis 7: Comparison: AZD7594 50 μg vs Placebo to AZD7594; Week 4; Test type: Superiority; p = 0.329, Mixed Models Analysis; Mean Difference (Final Values) = 0.931, 95% CI 2-sided [0.805 to 1.076]
Statistical Analysis 8: Comparison: AZD7594 90 μg vs Placebo to AZD7594; Week 4; Test type: Superiority; p = 0.203, Mixed Models Analysis; Mean Difference (Final Values) = 0.911, 95% CI 2-sided [0.789 to 1.052]
Statistical Analysis 9: Comparison: AZD7594 180 μg vs Placebo to AZD7594; Week 4; Test type: Superiority; p = 0.273, Mixed Models Analysis; Mean Difference (Final Values) = 0.923, 95% CI 2-sided [0.800 to 1.065]
Statistical Analysis 10: Comparison: AZD7594 360 μg vs Placebo to AZD7594; Week 4; Test type: Superiority; p = 0.023, Mixed Models Analysis; Mean Difference (Final Values) = 0.846, 95% CI 2-sided [0.734 to 0.977]
Statistical Analysis 11: Comparison: AZD7594 720 μg vs Placebo to AZD7594; Week 4; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.742, 95% CI 2-sided [0.646 to 0.852]
Statistical Analysis 12: Comparison: Placebo to AZD7594 vs Fluticasone Furoate; Week 4; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.703, 95% CI 2-sided [0.609 to 0.810]
Statistical Analysis 13: Comparison: AZD7594 50 μg vs Placebo to AZD7594; Week 8; Test type: Superiority; p = 0.283, Mixed Models Analysis; Mean Difference (Final Values) = 0.917, 95% CI 2-sided [0.783 to 1.074]
Statistical Analysis 14: Comparison: AZD7594 90 μg vs Placebo to AZD7594; Week 8; Test type: Superiority; p = 0.386, Mixed Models Analysis; Mean Difference (Final Values) = 0.933, 95% CI 2-sided [0.797 to 1.092]
Statistical Analysis 15: Comparison: AZD7594 180 μg vs Placebo to AZD7594; Week 8; Test type: Superiority; p = 0.126, Mixed Models Analysis; Mean Difference (Final Values) = 0.886, 95% CI 2-sided [0.758 to 1.035]
Statistical Analysis 16: Comparison: AZD7594 360 μg vs Placebo to AZD7594; Week 8; Test type: Superiority; p = 0.050, Mixed Models Analysis; Mean Difference (Final Values) = 0.855, 95% CI 2-sided [0.731 to 1.000]
Statistical Analysis 17: Comparison: AZD7594 720 μg vs Placebo to AZD7594; Week 8; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.723, 95% CI 2-sided [0.623 to 0.840]
Statistical Analysis 18: Comparison: Placebo to AZD7594 vs Fluticasone Furoate; Week 8; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.642, 95% CI 2-sided [0.550 to 0.749]
Statistical Analysis 19: Comparison: AZD7594 50 μg vs Placebo to AZD7594; Week 12; Test type: Superiority; p = 0.359, Mixed Models Analysis; Mean Difference (Final Values) = 0.927, 95% CI 2-sided [0.789 to 1.090]
Statistical Analysis 20: Comparison: AZD7594 90 μg vs Placebo to AZD7594; Week 12; Test type: Superiority; p = 0.556, Mixed Models Analysis; Mean Difference (Final Values) = 0.953, 95% CI 2-sided [0.813 to 1.118]
Statistical Analysis 21: Comparison: AZD7594 180 μg vs Placebo to AZD7594; Week 12; Test type: Superiority; p = 0.084, Mixed Models Analysis; Mean Difference (Final Values) = 0.869, 95% CI 2-sided [0.742 to 1.019]
Statistical Analysis 22: Comparison: AZD7594 360 μg vs Placebo to AZD7594; Week 12; Test type: Superiority; p = 0.011, Mixed Models Analysis; Mean Difference (Final Values) = 0.813, 95% CI 2-sided [0.693 to 0.953]
Statistical Analysis 23: Comparison: AZD7594 720 μg vs Placebo to AZD7594; Week 12; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.650, 95% CI 2-sided [0.559 to 0.757]
Statistical Analysis 24: Comparison: Placebo to AZD7594 vs Fluticasone Furoate; Week 12; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.623, 95% CI 2-sided [0.533 to 0.729]
Statistical Analysis 25: Comparison: AZD7594 50 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.231, Mixed Models Analysis; Mean Difference (Final Values) = 0.928, 95% CI 2-sided [0.821 to 1.049]
Statistical Analysis 26: Comparison: AZD7594 90 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.170, Mixed Models Analysis; Mean Difference (Final Values) = 0.918, 95% CI 2-sided [0.812 to 1.037]
Statistical Analysis 27: Comparison: AZD7594 180 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.039, Mixed Models Analysis; Mean Difference (Final Values) = 0.879, 95% CI 2-sided [0.778 to 0.994]
Statistical Analysis 28: Comparison: AZD7594 360 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.004, Mixed Models Analysis; Mean Difference (Final Values) = 0.835, 95% CI 2-sided [0.739 to 0.943]
Statistical Analysis 29: Comparison: AZD7594 720 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.700, 95% CI 2-sided [0.622 to 0.787]
Statistical Analysis 30: Comparison: Placebo to AZD7594 vs Fluticasone Furoate; Treatment period average; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.649, 95% CI 2-sided [0.575 to 0.732]

4. Secondary Outcome: Change From Baseline in Trough Forced Vital Capacity (FVC) at Week 12 and Average Over the Treatment Period
Description: Trough value was defined as the mean of the 2 measurements 30 minutes apart (23 hours after last dose) pre-dose for every visit throughout the Treatment Period (Visit 4/Week 2 to Visit 7/Week 12). Baseline was defined as the mean of the 2 measured values before first IP administration (30 minutes apart, at -45 minutes and -15 minutes, before IP administration) on Day 1 (Visit 3). Analyses were based on a MMRM with treatment, visit, treatment by visit interaction and region as fixed effects, and baseline value and baseline by visit interaction as covariates.
Time Frame: At week 12
Population: Full Analysis Set: All participants randomised and receiving at least 1 dose of randomised study drug.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | AZD7594 50 μg | AZD7594 90 μg | AZD7594 180 μg | AZD7594 360 μg | AZD7594 720 μg | Placebo to AZD7594 | Fluticasone Furoate
Number analyzed (Participants) | 110 | 112 | 111 | 113 | 134 | 113 | 112
Liters
  Week 12: number analyzed (Participants) | 83 | 90 | 92 | 90 | 123 | 70 | 103
  Week 12 | 0.027 [-0.047 to 0.101] | -0.017 [-0.089 to 0.056] | 0.076 [0.005 to 0.148] | 0.119 [0.047 to 0.191] | 0.088 [0.021 to 0.155] | 0.061 [-0.018 to 0.141] | 0.118 [0.048 to 0.188]
  Treatment Period Avg: number analyzed (Participants) | 108 | 109 | 108 | 109 | 132 | 95 | 110
  Treatment Period Avg | 0.044 [-0.017 to 0.106] | 0.019 [-0.041 to 0.080] | 0.087 [0.026 to 0.148] | 0.127 [0.066 to 0.188] | 0.091 [0.033 to 0.149] | 0.046 [-0.020 to 0.112] | 0.121 [0.062 to 0.181]
Statistical Analysis 1: Comparison: AZD7594 50 μg vs Placebo to AZD7594; Week 12; Test type: Superiority; p = 0.519, Mixed Models Analysis; Mean Difference (Final Values) = -0.034, 95% CI 2-sided [-0.139 to 0.070]
Statistical Analysis 2: Comparison: AZD7594 90 μg vs Placebo to AZD7594; Week 12; Test type: Superiority; p = 0.141, Mixed Models Analysis; Mean Difference (Final Values) = -0.078, 95% CI 2-sided [-0.181 to 0.026]
Statistical Analysis 3: Comparison: AZD7594 180 μg vs Placebo to AZD7594; Week 12; Test type: Superiority; p = 0.772, Mixed Models Analysis; Mean Difference (Final Values) = 0.015, 95% CI 2-sided [-0.088 to 0.119]
Statistical Analysis 4: Comparison: AZD7594 360 μg vs Placebo to AZD7594; Week 12; Test type: Superiority; p = 0.270, Mixed Models Analysis; Mean Difference (Final Values) = 0.058, 95% CI 2-sided [-0.045 to 0.162]
Statistical Analysis 5: Comparison: AZD7594 720 μg vs Placebo to AZD7594; Week 12; Test type: Superiority; p = 0.592, Mixed Models Analysis; Mean Difference (Final Values) = 0.027, 95% CI 2-sided [-0.072 to 0.126]
Statistical Analysis 6: Comparison: Placebo to AZD7594 vs Fluticasone Furoate; Week 12; Test type: Superiority; p = 0.275, Mixed Models Analysis; Mean Difference (Final Values) = 0.057, 95% CI 2-sided [-0.045 to 0.158]
Statistical Analysis 7: Comparison: AZD7594 50 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.963, Mixed Models Analysis; Mean Difference (Final Values) = -0.002, 95% CI 2-sided [-0.087 to 0.083]
Statistical Analysis 8: Comparison: AZD7594 90 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.533, Mixed Models Analysis; Mean Difference (Final Values) = -0.027, 95% CI 2-sided [-0.112 to 0.058]
Statistical Analysis 9: Comparison: AZD7594 180 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.342, Mixed Models Analysis; Mean Difference (Final Values) = 0.041, 95% CI 2-sided [-0.044 to 0.126]
Statistical Analysis 10: Comparison: AZD7594 360 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.061, Mixed Models Analysis; Mean Difference (Final Values) = 0.081, 95% CI 2-sided [-0.004 to 0.165]
Statistical Analysis 11: Comparison: AZD7594 720 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.278, Mixed Models Analysis; Mean Difference (Final Values) = 0.045, 95% CI 2-sided [-0.037 to 0.127]
Statistical Analysis 12: Comparison: Placebo to AZD7594 vs Fluticasone Furoate; Treatment period average; Test type: Superiority; p = 0.079, Mixed Models Analysis; Mean Difference (Final Values) = 0.075, 95% CI 2-sided [-0.009 to 0.159]

5. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire -5 (ACQ-5) at Week 12 and Average Over the Treatment Period
Description: Baseline was defined as the ACQ-5 score at Visit 3. Analyses were based on a MMRM with treatment, visit, treatment by visit interaction and region as fixed effects, and baseline value and baseline by visit interaction as covariates. To investigate the clinical efficacy of AZD7594 at different dose levels in asthmatics symptomatic on low dose ICS. Patients are asked to recall how their asthma was during the previous week and to evaluate their symptoms. The questionnaire has 5 items each item is scored on a scale of 0 to 6, where higher scores represent more severe impairment/symptoms. ACQ is the sum of the scores from all 5 items.
Time Frame: At week 12
Population: Full Analysis Set: All participants randomised and receiving at least 1 dose of randomised study drug.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | AZD7594 50 μg | AZD7594 90 μg | AZD7594 180 μg | AZD7594 360 μg | AZD7594 720 μg | Placebo to AZD7594 | Fluticasone Furoate
Number analyzed (Participants) | 110 | 112 | 111 | 113 | 134 | 113 | 112
units on a scale
  Week 12: number analyzed (Participants) | 83 | 91 | 93 | 90 | 122 | 70 | 103
  Week 12 | -0.289 [-0.412 to -0.166] | -0.394 [-0.513 to -0.274] | -0.357 [-0.476 to -0.239] | -0.330 [-0.449 to -0.210] | -0.406 [-0.514 to -0.297] | -0.137 [-0.269 to -0.004] | -0.360 [-0.474 to -0.245]
  Treatment Period Avg: number analyzed (Participants) | 108 | 110 | 108 | 110 | 132 | 101 | 110
  Treatment Period Avg | -0.215 [-0.307 to -0.122] | -0.230 [-0.322 to -0.139] | -0.220 [-0.311 to -0.128] | -0.291 [-0.382 to -0.199] | -0.306 [-0.394 to -0.219] | -0.090 [-0.187 to 0.008] | -0.269 [-0.359 to -0.179]
Statistical Analysis 1: Comparison: AZD7594 50 μg vs Placebo to AZD7594; Week 12; Test type: Superiority; p = 0.088, Mixed Models Analysis; Mean Difference (Final Values) = -0.153, 95% CI 2-sided [-0.328 to 0.023]
Statistical Analysis 2: Comparison: AZD7594 90 μg vs Placebo to AZD7594; Week 12; Test type: Superiority; p = 0.004, Mixed Models Analysis; Mean Difference (Final Values) = -0.257, 95% CI 2-sided [-0.430 to -0.084]
Statistical Analysis 3: Comparison: AZD7594 180 μg vs Placebo to AZD7594; Week 12; Test type: Superiority; p = 0.012, Mixed Models Analysis; Mean Difference (Final Values) = -0.221, 95% CI 2-sided [-0.393 to -0.049]
Statistical Analysis 4: Comparison: AZD7594 360 μg vs Placebo to AZD7594; Week 12; Test type: Superiority; p = 0.029, Mixed Models Analysis; Mean Difference (Final Values) = -0.193, 95% CI 2-sided [-0.366 to -0.020]
Statistical Analysis 5: Comparison: AZD7594 720 μg vs Placebo to AZD7594; Week 12; Test type: Superiority; p = 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.269, 95% CI 2-sided [-0.434 to -0.104]
Statistical Analysis 6: Comparison: Placebo to AZD7594 vs Fluticasone Furoate; Week 12; Test type: Superiority; p = 0.010, Mixed Models Analysis; Mean Difference (Final Values) = -0.223, 95% CI 2-sided [-0.393 to -0.054]
Statistical Analysis 7: Comparison: AZD7594 50 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.055, Mixed Models Analysis; Mean Difference (Final Values) = -0.125, 95% CI 2-sided [-0.253 to 0.003]
Statistical Analysis 8: Comparison: AZD7594 90 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.029, Mixed Models Analysis; Mean Difference (Final Values) = -0.141, 95% CI 2-sided [-0.268 to -0.014]
Statistical Analysis 9: Comparison: AZD7594 180 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.044, Mixed Models Analysis; Mean Difference (Final Values) = -0.130, 95% CI 2-sided [-0.257 to -0.003]
Statistical Analysis 10: Comparison: AZD7594 360 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.002, Mixed Models Analysis; Mean Difference (Final Values) = -0.201, 95% CI 2-sided [-0.328 to -0.074]
Statistical Analysis 11: Comparison: AZD7594 720 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.217, 95% CI 2-sided [-0.339 to -0.094]
Statistical Analysis 12: Comparison: Placebo to AZD7594 vs Fluticasone Furoate; Treatment period average; Test type: Superiority; p = 0.005, Mixed Models Analysis; Mean Difference (Final Values) = -0.179, 95% CI 2-sided [-0.305 to -0.053]

6. Secondary Outcome: Change From Baseline in Average Morning Peak Expiratory Flow (PEF) Over the Treatment Period
Description: Baseline was defined as the average over the 7 days prior to randomisation. Analyses were based on an ANCOVA model with treatment and region as fixed effects, and baseline value as a covariate. To investigate the clinical efficacy of AZD7594 at different dose levels in asthmatics symptomatic on low dose ICS.
Time Frame: Week 0 (7 days prior to randomisation) to Week 12
Population: Full Analysis Set: All participants randomised and receiving at least 1 dose of randomised study drug.
Measure: Least Squares Mean (95% Confidence Interval); unit: L/min
Arm/Group | AZD7594 50 μg | AZD7594 90 μg | AZD7594 180 μg | AZD7594 360 μg | AZD7594 720 μg | Placebo to AZD7594 | Fluticasone Furoate
Number analyzed (Participants) | 110 | 112 | 111 | 113 | 134 | 113 | 112
L/min | -4.036 [-10.518 to 2.447] | -5.718 [-11.994 to 0.557] | -2.576 [-8.768 to 3.617] | 3.745 [-2.558 to 10.048] | 4.900 [-1.010 to 10.810] | -11.699 [-18.749 to -4.649] | -1.208 [-7.209 to 4.793]
Statistical Analysis 1: Comparison: AZD7594 50 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.097, Mixed Models Analysis; Mean Difference (Final Values) = 7.664, 95% CI 2-sided [-1.403 to 16.730]
Statistical Analysis 2: Comparison: AZD7594 90 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.190, Mixed Models Analysis; Mean Difference (Final Values) = 5.981, 95% CI 2-sided [-2.980 to 14.941]
Statistical Analysis 3: Comparison: AZD7594 180 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.045, Mixed Models Analysis; Mean Difference (Final Values) = 9.123, 95% CI 2-sided [0.195 to 18.052]
Statistical Analysis 4: Comparison: AZD7594 360 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 15.444, 95% CI 2-sided [6.443 to 24.445]
Statistical Analysis 5: Comparison: AZD7594 720 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 16.599, 95% CI 2-sided [8.031 to 25.167]
Statistical Analysis 6: Comparison: Placebo to AZD7594 vs Fluticasone Furoate; Treatment period average; Test type: Superiority; p = 0.019, Mixed Models Analysis; Mean Difference (Final Values) = 10.491, 95% CI 2-sided [1.726 to 19.256]

7. Secondary Outcome: Change From Baseline in Average Evening PEF Over the Treatment Period
Description: as for outcome 6
Time Frame: Week 0 (7 days prior to randomisation) to Week 12
Population: Full Analysis set: All participants randomised and receiving at least 1 dose of randomised study drug.
Measure: Least Squares Mean (95% Confidence Interval); unit: L/min
Arm/Group | AZD7594 50 μg | AZD7594 90 μg | AZD7594 180 μg | AZD7594 360 μg | AZD7594 720 μg | Placebo to AZD7594 | Fluticasone Furoate
Number analyzed (Participants) | 110 | 112 | 111 | 113 | 134 | 113 | 112
L/min | -5.418 [-11.792 to 0.955] | -5.654 [-11.843 to 0.534] | -3.983 [-10.081 to 2.114] | 2.441 [-3.738 to 8.620] | 4.178 [-1.642 to 9.997] | -7.816 [-14.712 to -0.921] | -1.687 [-7.602 to 4.227]
Statistical Analysis 1: Comparison: AZD7594 50 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.597, Mixed Models Analysis; Mean Difference (Final Values) = 2.398, 95% CI 2-sided [-6.494 to 11.290]
Statistical Analysis 2: Comparison: AZD7594 90 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.629, Mixed Models Analysis; Mean Difference (Final Values) = 2.162, 95% CI 2-sided [-6.623 to 10.948]
Statistical Analysis 3: Comparison: AZD7594 180 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.389, Mixed Models Analysis; Mean Difference (Final Values) = 3.833, 95% CI 2-sided [-4.907 to 12.573]
Statistical Analysis 4: Comparison: AZD7594 360 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.022, Mixed Models Analysis; Mean Difference (Final Values) = 10.258, 95% CI 2-sided [1.456 to 19.059]
Statistical Analysis 5: Comparison: AZD7594 720 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.005, Mixed Models Analysis; Mean Difference (Final Values) = 11.994, 95% CI 2-sided [3.571 to 20.417]
Statistical Analysis 6: Comparison: Placebo to AZD7594 vs Fluticasone Furoate; Treatment period average; Test type: Superiority; p = 0.163, Mixed Models Analysis; Mean Difference (Final Values) = 6.129, 95% CI 2-sided [-2.479 to 14.737]

8. Secondary Outcome: Change From Baseline in Average Daily Use of Rescue Medication Over the Treatment Period
Description: To investigate the clinical efficacy of AZD7594 at different dose levels in asthmatics symptomatic on low dose ICS. Baseline was defined as the average over the 7 days prior to randomisation. Analyses were based on an ANCOVA model with treatment and region as fixed effects, and baseline value as a covariate.
Time Frame: Week 0 (7 days prior to randomisation) to Week 12
Population: Full Analysis Set: All participants randomised and receiving at least 1 dose of randomised study drug.
Measure: Least Squares Mean (95% Confidence Interval); unit: number of puffs
Arm/Group | AZD7594 50 μg | AZD7594 90 μg | AZD7594 180 μg | AZD7594 360 μg | AZD7594 720 μg | Placebo to AZD7594 | Fluticasone Furoate
Number analyzed (Participants) | 110 | 112 | 111 | 113 | 134 | 113 | 112
number of puffs | -0.370 [-0.502 to -0.237] | -0.282 [-0.415 to -0.149] | -0.226 [-0.356 to -0.096] | -0.435 [-0.572 to -0.297] | -0.435 [-0.560 to -0.310] | -0.127 [-0.276 to 0.023] | -0.304 [-0.432 to -0.175]
Statistical Analysis 1: Comparison: AZD7594 50 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.012, Mixed Models Analysis; Mean Difference (Final Values) = -0.243, 95% CI 2-sided [-0.431 to -0.054]
Statistical Analysis 2: Comparison: AZD7594 90 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.108, Mixed Models Analysis; Mean Difference (Final Values) = -0.155, 95% CI 2-sided [-0.344 to 0.034]
Statistical Analysis 3: Comparison: AZD7594 180 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.295, Mixed Models Analysis; Mean Difference (Final Values) = -0.099, 95% CI 2-sided [-0.286 to 0.087]
Statistical Analysis 4: Comparison: AZD7594 360 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.002, Mixed Models Analysis; Mean Difference (Final Values) = -0.308, 95% CI 2-sided [-0.500 to -0.116]
Statistical Analysis 5: Comparison: AZD7594 720 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.308, 95% CI 2-sided [-0.489 to -0.126]
Statistical Analysis 6: Comparison: Placebo to AZD7594 vs Fluticasone Furoate; Treatment period average; Test type: Superiority; p = 0.062, Mixed Models Analysis; Mean Difference (Final Values) = -0.177, 95% CI 2-sided [-0.362 to 0.009]

9. Secondary Outcome: Change From Baseline in Percent Night-time Awakening Days Over the Treatment Period
Description: as for outcome 8
Time Frame: Week 0 (7 days prior to randomisation) to Week 12
Population: Full Analysis Set: All participants randomised and receiving at least 1 dose of randomised study drug.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage
Arm/Group | AZD7594 50 μg | AZD7594 90 μg | AZD7594 180 μg | AZD7594 360 μg | AZD7594 720 μg | Placebo to AZD7594 | Fluticasone Furoate
Number analyzed (Participants) | 110 | 112 | 111 | 113 | 134 | 113 | 112
percentage | -14.281 [-18.408 to -10.154] | -12.260 [-16.263 to -8.257] | -8.649 [-12.579 to -4.718] | -12.085 [-16.102 to -8.068] | -13.017 [-16.790 to -9.244] | -4.288 [-8.814 to 0.238] | -15.910 [-19.753 to -12.067]
Statistical Analysis 1: Comparison: AZD7594 50 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -9.993, 95% CI 2-sided [-15.795 to -4.191]
Statistical Analysis 2: Comparison: AZD7594 90 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.006, Mixed Models Analysis; Mean Difference (Final Values) = -7.972, 95% CI 2-sided [-13.694 to -2.251]
Statistical Analysis 3: Comparison: AZD7594 180 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.133, Mixed Models Analysis; Mean Difference (Final Values) = -4.361, 95% CI 2-sided [-10.051 to 1.329]
Statistical Analysis 4: Comparison: AZD7594 360 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.008, Mixed Models Analysis; Mean Difference (Final Values) = -7.797, 95% CI 2-sided [-13.555 to -2.040]
Statistical Analysis 5: Comparison: AZD7594 720 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.002, Mixed Models Analysis; Mean Difference (Final Values) = -8.729, 95% CI 2-sided [-14.195 to -3.264]
Statistical Analysis 6: Comparison: Placebo to AZD7594 vs Fluticasone Furoate; Treatment period average; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -11.622, 95% CI 2-sided [-17.211 to -6.034]

10. Secondary Outcome: Change From Baseline in Average Daily Asthma Symptom Score Over the Treatment Period
Description: To investigate the clinical efficacy of AZD7594 at different dose levels in asthmatics symptomatic on low dose ICS (Full Analysis Set). Baseline was defined as the average over the 7 days prior to randomisation. Analyses were based on an ANCOVA model with treatment and region as fixed effects, and baseline value as a covariate. During the Run-in and Treatment Periods, subjects recorded the severity of their asthma symptoms during night-time and day-time each morning and evening, using the eDiary. Asthma symptom scores during night-time/day-time were assessed by the subject each morning/evening according to the following scoring system and recorded on the eDiary: 0: No asthma symptoms, 1: The subjects were aware of their asthma symptoms but they can easily tolerate the symptoms, 2: asthma was causing enough discomfort to cause problems with sleep, 3: Subjects were unable to sleep/do normal activities because of their asthma.
Time Frame: Week 0 (7 days prior to randomisation) to Week 12
Population: Full Analysis Set: All participants randomised and receiving at least 1 dose of randomised study drug.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | AZD7594 50 μg | AZD7594 90 μg | AZD7594 180 μg | AZD7594 360 μg | AZD7594 720 μg | Placebo to AZD7594 | Fluticasone Furoate
Number analyzed (Participants) | 110 | 112 | 111 | 113 | 134 | 113 | 112
units on a scale | -0.303 [-0.385 to -0.220] | -0.201 [-0.283 to -0.118] | -0.229 [-0.310 to -0.149] | -0.321 [-0.407 to -0.235] | -0.275 [-0.353 to -0.198] | -0.091 [-0.184 to 0.003] | -0.296 [-0.376 to -0.216]
Statistical Analysis 1: Comparison: AZD7594 50 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.212, 95% CI 2-sided [-0.329 to -0.094]
Statistical Analysis 2: Comparison: AZD7594 90 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.066, Mixed Models Analysis; Mean Difference (Final Values) = -0.110, 95% CI 2-sided [-0.228 to 0.007]
Statistical Analysis 3: Comparison: AZD7594 180 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.020, Mixed Models Analysis; Mean Difference (Final Values) = -0.139, 95% CI 2-sided [-0.255 to -0.022]
Statistical Analysis 4: Comparison: AZD7594 360 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.230, 95% CI 2-sided [-0.350 to -0.110]
Statistical Analysis 5: Comparison: AZD7594 720 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.185, 95% CI 2-sided [-0.298 to -0.071]
Statistical Analysis 6: Comparison: Placebo to AZD7594 vs Fluticasone Furoate; Treatment period average; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.206, 95% CI 2-sided [-0.321 to -0.090]

11. Secondary Outcome: Change From Baseline in Percent Asthma Control Days Over the Treatment Period
Description: To investigate the clinical efficacy of AZD7594 at different dose levels in asthmatics symptomatic on low dose ICS. Asthma-control days is defined as days with no symptoms, nonight-waking, no reliever use, and no exacerbation. Baseline was defined as the average over the 7 days prior to randomisation. Analyses were based on an ANCOVA model with treatment and region as fixed effects, and baseline value as a covariate.
Time Frame: Week 0 (7 days prior to randomisation) to Week 12
Population: Full Analysis Set: All participants randomised and receiving at least 1 dose of randomised study drug.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent
Arm/Group | AZD7594 50 μg | AZD7594 90 μg | AZD7594 180 μg | AZD7594 360 μg | AZD7594 720 μg | Placebo to AZD7594 | Fluticasone Furoate
Number analyzed (Participants) | 110 | 112 | 111 | 113 | 134 | 113 | 112
percent | 15.470 [9.547 to 21.394] | 11.362 [5.435 to 17.290] | 12.646 [6.865 to 18.427] | 15.925 [9.775 to 22.076] | 14.479 [8.896 to 20.062] | 5.859 [-0.813 to 12.532] | 13.037 [7.301 to 18.772]
Statistical Analysis 1: Comparison: AZD7594 50 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.026, Mixed Models Analysis; Mean Difference (Final Values) = 9.611, 95% CI 2-sided [1.180 to 18.042]
Statistical Analysis 2: Comparison: AZD7594 90 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.200, Mixed Models Analysis; Mean Difference (Final Values) = 5.503, 95% CI 2-sided [-2.927 to 13.933]
Statistical Analysis 3: Comparison: AZD7594 180 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.110, Mixed Models Analysis; Mean Difference (Final Values) = 6.787, 95% CI 2-sided [-1.546 to 15.119]
Statistical Analysis 4: Comparison: AZD7594 360 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.022, Mixed Models Analysis; Mean Difference (Final Values) = 10.066, 95% CI 2-sided [1.461 to 18.672]
Statistical Analysis 5: Comparison: AZD7594 720 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.038, Mixed Models Analysis; Mean Difference (Final Values) = 8.620, 95% CI 2-sided [0.489 to 16.750]
Statistical Analysis 6: Comparison: Placebo to AZD7594 vs Fluticasone Furoate; Treatment period average; Test type: Superiority; p = 0.090, Mixed Models Analysis; Mean Difference (Final Values) = 7.178, 95% CI 2-sided [-1.112 to 15.467]

12. Secondary Outcome: Change From Baseline in Percent Rescue-free Days Over the Treatment Period
Description: To investigate the clinical efficacy of AZD7594 at different dose levels in asthmatics symptomatic on low dose ICS. A rescue-free day (RFD) was defined as a day where the number of puffs of medication for the relief of asthma symptoms was reported as zero. Baseline was defined as the average over the 7 days prior to randomisation. Analyses were based on an ANCOVA model with treatment and region as fixed effects, and baseline value as a covariate.
Time Frame: Week 0 (7 days prior to randomisation) to Week 12
Population: Full Analysis Set: All participants randomised and receiving at least 1 dose of randomised study drug.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent
Arm/Group | AZD7594 50 μg | AZD7594 90 μg | AZD7594 180 μg | AZD7594 360 μg | AZD7594 720 μg | Placebo to AZD7594 | Fluticasone Furoate
Number analyzed (Participants) | 110 | 112 | 111 | 113 | 134 | 113 | 112
percent | 31.138 [24.019 to 38.257] | 24.178 [17.045 to 31.312] | 21.960 [14.940 to 28.980] | 34.991 [27.549 to 42.433] | 30.775 [24.025 to 37.526] | 23.202 [15.188 to 31.215] | 28.260 [21.308 to 35.211]
Statistical Analysis 1: Comparison: AZD7594 50 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.123, Mixed Models Analysis; Mean Difference (Final Values) = 7.936, 95% CI 2-sided [-2.160 to 18.031]
Statistical Analysis 2: Comparison: AZD7594 90 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.849, Mixed Models Analysis; Mean Difference (Final Values) = 0.977, 95% CI 2-sided [-9.112 to 11.065]
Statistical Analysis 3: Comparison: AZD7594 180 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.807, Mixed Models Analysis; Mean Difference (Final Values) = -1.242, 95% CI 2-sided [-11.233 to 8.748]
Statistical Analysis 4: Comparison: AZD7594 360 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.025, Mixed Models Analysis; Mean Difference (Final Values) = 11.789, 95% CI 2-sided [1.488 to 22.090]
Statistical Analysis 5: Comparison: AZD7594 720 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.127, Mixed Models Analysis; Mean Difference (Final Values) = 7.574, 95% CI 2-sided [-2.160 to 17.307]
Statistical Analysis 6: Comparison: Placebo to AZD7594 vs Fluticasone Furoate; Treatment period average; Test type: Superiority; p = 0.318, Mixed Models Analysis; Mean Difference (Final Values) = 5.058, 95% CI 2-sided [-4.874 to 14.990]

13. Secondary Outcome: Change From Baseline in Percent Symptom-free Days Over the Treatment Period
Description: To investigate the clinical efficacy of AZD7594 at different dose levels in asthmatics symptomatic on low dose ICS. Days without asthma symptoms, or symptom-free days, are defined as a day without asthma symptoms, short-acting β-agonist (SABA) use, systemic corticosteroid use, or need for urgent asthma care.
Time Frame: Week 0 (7 days prior to randomisation) to Week 12
Population: Full Analysis Set: All participants randomised and receiving at least 1 dose of randomised study drug.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent
Arm/Group | AZD7594 50 μg | AZD7594 90 μg | AZD7594 180 μg | AZD7594 360 μg | AZD7594 720 μg | Placebo to AZD7594 | Fluticasone Furoate
Number analyzed (Participants) | 110 | 112 | 111 | 113 | 134 | 113 | 112
percent | 13.780 [7.873 to 19.686] | 10.521 [4.608 to 16.435] | 11.935 [6.169 to 17.701] | 14.673 [8.539 to 20.806] | 13.451 [7.883 to 19.018] | 3.329 [-3.319 to 9.977] | 14.018 [8.293 to 19.743]
Statistical Analysis 1: Comparison: AZD7594 50 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.015, Mixed Models Analysis; Mean Difference (Final Values) = 10.450, 95% CI 2-sided [2.046 to 18.855]
Statistical Analysis 2: Comparison: AZD7594 90 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.093, Mixed Models Analysis; Mean Difference (Final Values) = 7.192, 95% CI 2-sided [-1.208 to 15.592]
Statistical Analysis 3: Comparison: AZD7594 180 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.042, Mixed Models Analysis; Mean Difference (Final Values) = 8.606, 95% CI 2-sided [0.298 to 16.913]
Statistical Analysis 4: Comparison: AZD7594 360 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.010, Mixed Models Analysis; Mean Difference (Final Values) = 11.344, 95% CI 2-sided [2.773 to 19.914]
Statistical Analysis 5: Comparison: AZD7594 720 μg vs Placebo to AZD7594; Treatment period average; Test type: Superiority; p = 0.014, Mixed Models Analysis; Mean Difference (Final Values) = 10.122, 95% CI 2-sided [2.021 to 18.222]
Statistical Analysis 6: Comparison: Placebo to AZD7594 vs Fluticasone Furoate; Treatment period average; Test type: Superiority; p = 0.011, Mixed Models Analysis; Mean Difference (Final Values) = 10.689, 95% CI 2-sided [2.424 to 18.953]

14. Secondary Outcome: Observed Maximum Concentration at Steady State (Css,Max) of AZD7594 at Day 84
Description: Summary of PK parameter Css,mx, observed maximum concentration, of AZD7594 at day 84 in PK analysis set. The presented results are summary statistics of the PK parameter.
Time Frame: Day 84 (pre-dose and 0.25, 0.5, 1.0, 2.0, 4.0, 8.0, 12.0, 16.0 and 24 h post-dose)
Population: All randomised patients participating in the PK subset, who took at least one dose of IP and for whom at least one of the primary PK parameters could be calculated, and who had no major protocol deviations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol/L
Arm/Group | AZD7594 50 μg | AZD7594 90 μg | AZD7594 180 μg | AZD7594 360 μg | AZD7594 720 μg | Placebo to AZD7594 | Fluticasone Furoate
Number analyzed (Participants) | 18 | 14 | 16 | 16 | 28 | 0 | 0
pmol/L | 48.45 (68.65) | 114.90 (99.12) | 69.71 (105.94) | 154.50 (144.67) | 200.00 (113.05) |  |

15. Secondary Outcome: Observed Minimum Concentration at the End of the Dosing Interval (Css,Min) of AZD7594 at Day 84
Description: Summary of PK parameter Css,min, observed minimum concentration, of AZD7594 at day 84 in PK analysis set. The presented results are summary statistics of the PK parameter.
Time Frame: Day 84 (pre-dose and 0.25, 0.5, 1.0, 2.0, 4.0, 8.0, 12.0, 16.0 and 24 h post-dose)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol/L
Arm/Group | AZD7594 50 μg | AZD7594 90 μg | AZD7594 180 μg | AZD7594 360 μg | AZD7594 720 μg | Placebo to AZD7594 | Fluticasone Furoate
Number analyzed (Participants) | 18 | 14 | 16 | 16 | 28 | 0 | 0
pmol/L | 14.41 (37.59) | 21.45 (43.12) | 30.22 (43.28) | 70.58 (46.22) | 85.13 (108.41) |  |

16. Secondary Outcome: Time to Maximum Concentration at Steady State, Taken Directly From the Individual Concentration-time Curve (Tss, Max) of AZD7594 at Day 84
Description: Summary of PK parameter tss, max, Time to maximum concentration at steady state, taken directly from the individual concentration-time curve, of AZD7594 at day 84 in PK analysis set. The presented results are summary statistics of the PK parameter.
Time Frame: Day 84 (pre-dose and 0.25, 0.5, 1.0, 2.0, 4.0, 8.0, 12.0, 16.0 and 24 h post-dose)
Population: as for outcome 14
Measure: Median (Full Range); unit: hours
Arm/Group | AZD7594 50 μg | AZD7594 90 μg | AZD7594 180 μg | AZD7594 360 μg | AZD7594 720 μg | Placebo to AZD7594 | Fluticasone Furoate
Number analyzed (Participants) | 18 | 14 | 16 | 16 | 28 | 0 | 0
hours | 0.25 [0.23 to 2.17] | 0.25 [0.00 to 0.98] | 0.25 [0.20 to 2.00] | 0.25 [0.00 to 2.00] | 0.25 [0.00 to 23.98] |  |

17. Secondary Outcome: Time of Last Quantifiable Analyte Concentration (Tlast) of AZD7594 at Day 84
Description: Summary of PK parameter Tlast, Time of last quantifiable analyte concentration, of AZD7594 at day 84 in PK analysis set. The presented results are summary statistics of the PK parameter.
Time Frame: Day 84 (pre-dose and 0.25, 0.5, 1.0, 2.0, 4.0, 8.0, 12.0, 16.0 and 24 h post-dose)
Population: as for outcome 14
Measure: Median (Full Range); unit: hours
Arm/Group | AZD7594 50 μg | AZD7594 90 μg | AZD7594 180 μg | AZD7594 360 μg | AZD7594 720 μg | Placebo to AZD7594 | Fluticasone Furoate
Number analyzed (Participants) | 18 | 14 | 16 | 16 | 28 | 0 | 0
hours | 8.01 [0.50 to 24.07] | 24.00 [4.00 to 24.17] | 24.00 [0.25 to 24.05] | 24.00 [12.00 to 24.05] | 24.00 [23.92 to 24.03] |  |

18. Secondary Outcome: Area Under the Plasma Concentration-curve From Time Zero to the Time of Last Quantifiable Analyte Concentration (AUClast) of AZD7594 at Day 84
Description: Summary of PK parameter AUClast, Area under the plasma concentration-curve from time zero to the time of last quantifiable analyte concentration, of AZD7594 at day 84 in PK analysis set. The presented results are summary statistics of the PK parameter.
Time Frame: Day 84 (pre-dose and 0.25, 0.5, 1.0, 2.0, 4.0, 8.0, 12.0, 16.0 and 24 h post-dose)
Population: All randomized patients participating in the PK subset, who took at least one dose of IP and for whom at least one of the primary PK parameters could be calculated, and who had no major protocol deviations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pmol/L
Arm/Group | AZD7594 50 μg | AZD7594 90 μg | AZD7594 180 μg | AZD7594 360 μg | AZD7594 720 μg | Placebo to AZD7594 | Fluticasone Furoate
Number analyzed (Participants) | 18 | 14 | 16 | 16 | 28 | 0 | 0
h*pmol/L | 167.50 (123.50) | 573.00 (116.00) | 719.10 (134.58) | 1435.00 (140.28) | 2622.00 (98.88) |  |

19. Secondary Outcome: Area Under the Plasma Concentration-curve Within a Dosing Interval (AUCτ) of AZD7594 at Day 84
Description: Summary of PK parameter AUCτ, Area under the plasma concentration-curve within a dosing interval, of AZD7594 at day 84 in PK analysis set. The presented results are summary statistics of the PK parameter.
Time Frame: Day 84 (pre-dose and 0.25, 0.5, 1.0, 2.0, 4.0, 8.0, 12.0, 16.0 and 24 h post-dose)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pmol/L
Arm/Group | AZD7594 50 μg | AZD7594 90 μg | AZD7594 180 μg | AZD7594 360 μg | AZD7594 720 μg | Placebo to AZD7594 | Fluticasone Furoate
Number analyzed (Participants) | 18 | 14 | 16 | 16 | 28 | 0 | 0
h*pmol/L | 530.50 (32.57) | 928.60 (37.52) | 1137.00 (52.06) | 2205.00 (52.32) | 2622.00 (98.88) |  |

20. Secondary Outcome: Average Plasma Concentration During a Dosing Interval at Steady State (Css,Avg) of AZD7594 at Day 84
Description: Summary of PK parameter Css,avg, Average plasma concentration during a dosing interval at steady state, of AZD7594 at day 84 in PK analysis set. The presented results are summary statistics of the PK parameter.
Time Frame: Day 84 (pre-dose and 0.25, 0.5, 1.0, 2.0, 4.0, 8.0, 12.0, 16.0 and 24 h post-dose)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol/L
Arm/Group | AZD7594 50 μg | AZD7594 90 μg | AZD7594 180 μg | AZD7594 360 μg | AZD7594 720 μg | Placebo to AZD7594 | Fluticasone Furoate
Number analyzed (Participants) | 18 | 14 | 16 | 16 | 28 | 0 | 0
pmol/L | 22.10 (32.57) | 38.69 (37.52) | 47.37 (52.06) | 91.86 (52.32) | 109.30 (98.88) |  |

21. Secondary Outcome: Dose Normalised Css,Max (Css,Max/D) of AZD7594 at Day 84
Description: Summary of PK parameter Css,max/D Dose normalised Css,max, of AZD7594 at day 84 in PK analysis set. The presented results are summary statistics of the PK parameter.
Time Frame: Day 84 (pre-dose and 0.25, 0.5, 1.0, 2.0, 4.0, 8.0, 12.0, 16.0 and 24 h post-dose)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol/L/umol
Arm/Group | AZD7594 50 μg | AZD7594 90 μg | AZD7594 180 μg | AZD7594 360 μg | AZD7594 720 μg | Placebo to AZD7594 | Fluticasone Furoate
Number analyzed (Participants) | 18 | 14 | 16 | 16 | 28 | 0 | 0
pmol/L/umol | 587.80 (68.65) | 774.40 (99.12) | 234.90 (105.94) | 260.40 (144.67) | 168.50 (113.05) |  |

22. Secondary Outcome: Dose Normalised AUCτ (AUCτ/D) of AZD7594 at Day 84
Description: Summary of PK parameter AUCτ/D, Dose normalised AUCτ, of AZD7594 at day 84 in PK analysis set. The presented results are summary statistics of the PK parameter.
Time Frame: Day 84 (pre-dose and 0.25, 0.5, 1.0, 2.0, 4.0, 8.0, 12.0, 16.0 and 24 h post-dose)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pmol/μmol
Arm/Group | AZD7594 50 μg | AZD7594 90 μg | AZD7594 180 μg | AZD7594 360 μg | AZD7594 720 μg | Placebo to AZD7594 | Fluticasone Furoate
Number analyzed (Participants) | 18 | 14 | 16 | 16 | 28 | 0 | 0
h*pmol/μmol | 6436.00 (32.57) | 6259.00 (37.52) | 3831.00 (52.06) | 3715.00 (52.32) | 2209.00 (98.88) |  |

23. Secondary Outcome: Percentage Fluctuation of AZD7594 at Day 84
Description: To describe the (steady state) PK of AZD7594 in a subset of asthmatics symptomatic on low dose ICS (subset of subjects at EU sites) (PK Analysis Set). The presented results are summary statistics of the PK parameter. No statistical analysis is done for this endpoint. Fluctuation index during a dosing interval estimated as 100*(Css,max - Css,min)/Css,avg (%), where Css,min is the minimum concentration at the end of the dosing interval.
Time Frame: Day 84 (pre-dose and 0.25, 0.5, 1.0, 2.0, 4.0, 8.0, 12.0, 16.0 and 24 h post-dose)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage
Arm/Group | AZD7594 50 μg | AZD7594 90 μg | AZD7594 180 μg | AZD7594 360 μg | AZD7594 720 μg | Placebo to AZD7594 | Fluticasone Furoate
Number analyzed (Participants) | 18 | 14 | 16 | 16 | 28 | 0 | 0
percentage | 387.80 (21.97) | 326.60 (37.40) | 148.90 (38.27) | 172.10 (44.32) | 98.22 (61.36) |  |

24. Secondary Outcome: Change From Baseline in Area Under Plasma Cortisol Concentration-time Curve (AUEC0-24hrs Post Dose), of AZD7594 vs Placebo at Day 84
Description: Area under the plasma cortisol concentration-time curve from zero to 24 hours after dosing compared to Placebo, of AZD7594 at day 84 in PK analysis set. The presented results are summary statistics of the PK parameter.
Time Frame: At Day -1 (-24 to -12 h prior to the dose on Day 0) and at Day 84 (0 to 12 hours post dose)
Population: All randomised patients who took at least one dose of IP and for whom 24-hour cortisol sampling was performed and baseline and post baseline AUEC0-24 could be calculated.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ng*hr/mL
Arm/Group | AZD7594 50 μg | AZD7594 90 μg | AZD7594 180 μg | AZD7594 360 μg | AZD7594 720 μg | Placebo to AZD7594 | Fluticasone Furoate
Number analyzed (Participants) | 110 | 112 | 111 | 113 | 134 | 113 | 112
ng*hr/mL | 1.029 [0.920 to 1.152] | 1.140 [1.009 to 1.287] | 1.151 [1.018 to 1.300] | 1.003 [0.891 to 1.129] | 0.934 [0.850 to 1.026] | 1.019 [0.895 to 1.161] | 1.011 [0.898 to 1.137]
Statistical Analysis 1: Comparison: AZD7594 50 μg vs Placebo to AZD7594; Test type: Superiority; p = 0.909, Mixed Models Analysis; geometric LSMean ratio = 1.010, 95% CI 2-sided [0.851 to 1.199]
Statistical Analysis 2: Comparison: AZD7594 90 μg vs Placebo to AZD7594; Test type: Superiority; p = 0.218, Mixed Models Analysis; geometric LSMean ratio = 1.118, 95% CI 2-sided [0.935 to 1.336]
Statistical Analysis 3: Comparison: AZD7594 180 μg vs Placebo to AZD7594; Test type: Superiority; p = 0.181, Mixed Models Analysis; geometric LSMean ratio = 1.129, 95% CI 2-sided [0.944 to 1.349]
Statistical Analysis 4: Comparison: AZD7594 360 μg vs Placebo to AZD7594; Test type: Superiority; p = 0.859, Mixed Models Analysis; geometric LSMean ratio = 0.984, 95% CI 2-sided [0.825 to 1.174]
Statistical Analysis 5: Comparison: AZD7594 720 μg vs Placebo to AZD7594; Test type: Superiority; p = 0.285, Mixed Models Analysis; geometric LSMean ratio = 0.916, 95% CI 2-sided [0.780 to 1.077]
Statistical Analysis 6: Comparison: Placebo to AZD7594 vs Fluticasone Furoate; Test type: Superiority; p = 0.923, Mixed Models Analysis; geometric LSMean ratio = 0.991, 95% CI 2-sided [0.831 to 1.182]

25. Secondary Outcome: Number of Participants With Adverse Events
Description: To evaluate the safety and tolerability of AZD7594 in relation to Placebo in asthmatics symptomatic on low dose ICS
Time Frame: From screening to follow-up period (7 to 10 days after visit 7)
Population: All participants randomised and receiving at least 1 dose of randomised study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD7594 50 μg | AZD7594 90 μg | AZD7594 180 μg | AZD7594 360 μg | AZD7594 720 μg | Placebo to AZD7594 | Fluticasone Furoate
Number analyzed (Participants) | 110 | 112 | 111 | 113 | 134 | 113 | 112
Participants
  Any AE | 35 | 45 | 39 | 54 | 46 | 47 | 34
  death | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Any SAE | 0 | 3 | 1 | 3 | 3 | 0 | 1
  Any AE leading to discontinuation of IP | 6 | 8 | 4 | 11 | 4 | 20 | 2

ADVERSE EVENTS:
Time Frame: From Screening to follow-up period (7 to 10 days after visit 7), maximum up to 1 year.
Description: An AE was the development of an undesirable medical condition or the deterioration of a preexisting medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product. An undesirable medical condition could be symptoms (e.g: nausea, chest pain), signs (e.g: tachycardia, enlarged liver) or abnormal results of an investigation (e.g., laboratory findings, electrocardiogram). SAEs were recorded from the time of informed consent.
Arm/Group | AZD7594 50 μg | AZD7594 90 μg | AZD7594 180 μg | AZD7594 360 μg | AZD7594 720 μg | Placebo to AZD7594 | Fluticasone Furoate
All-Cause Mortality (participants affected / at risk) | 0/110 | 0/112 | 0/111 | 1/113 | 0/134 | 0/113 | 0/112
Serious Adverse Events (participants affected / at risk) | 0/110 | 3/112 | 1/111 | 3/113 | 3/134 | 0/113 | 1/112
Other Adverse Events (participants affected / at risk) | 14/110 | 15/112 | 8/111 | 14/113 | 8/134 | 24/113 | 11/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD7594 50 μg (N=110) | AZD7594 90 μg (N=112) | AZD7594 180 μg (N=111) | AZD7594 360 μg (N=113) | AZD7594 720 μg (N=134) | Placebo to AZD7594 (N=113) | Fluticasone Furoate (N=112)
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD7594 50 μg (N=110) | AZD7594 90 μg (N=112) | AZD7594 180 μg (N=111) | AZD7594 360 μg (N=113) | AZD7594 720 μg (N=134) | Placebo to AZD7594 (N=113) | Fluticasone Furoate (N=112)
Nasopharyngitis (Infections and infestations) | 7 | 9 | 6 | 4 | 5 | 6 | 9
Asthma (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 2 | 10 | 3 | 19 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-04-26): https://cdn.clinicaltrials.gov/large-docs/12/NCT03622112/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-30): https://cdn.clinicaltrials.gov/large-docs/12/NCT03622112/SAP_001.pdf